CLINICAL TRIAL: NCT03031444
Title: A Multicenter Study of Prognosis and the Efficacy Comparison of Perioperative Chemotherapy Plus Cetuximab Versus Chemotherapy Alone for High Risk Patients(Clinical Risk Score≥3) of Resectable Colorectal Liver Metastasis
Brief Title: Perioperative Chemotherapy Plus Cetuximab Versus Chemotherapy Alone for High Risk Resectable Colorectal Liver Metastasis
Acronym: PARECEC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Beijing Municipal Administration of Hospitals (Other Government); West China Hospital (Other); Zhejiang Cancer Hospital (Other); First Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Principal Investigator, Wang Kun, associate director, Peking University Cancer Hospital & Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PX2016002
Record Dates: First submitted 2016-12-04; First posted 2017-01-25 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Colorectal Cancer Stage IV; Metastasis
Keywords: colorectal liver metastasis; preoperative; chemotherapy; targeted therapy
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Cetuximab; Folfox protocol; XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- chemotherapy plus cetuximab (Active Comparator): Cetuximab plus FOLFIRI/FOLFOX:FOLFIRI plus cetuximab [Irinotecan 180 mg/m2 IV over 30-90 minutes, day 1;Leucovorin 400 mg/m2 IV infusion to match duration of irinotecan infusion, day 1;5-fluoruracil(5-FU) 400 mg/m2 IV bolus day 1, then 1200 mg/m2/day x 2 days (total 2400 mg/m2 over 46-48 hours) IV continuous infusion.Repeat every 2 weeks.Cetuximab 500 mg/m2 IV over 2 hours, day 1, every 2 weeks] or FOLFOX plus Cetuximab [Oxaliplatin 85 mg/m2 IV over 2 hours, day 1 Leucovorin 400 mg/m2 IV over 2 hours, day 1 5-FU 400 mg/m2 IV bolus on day 1, then 1200 mg/m2/day x 2 days (total 2400 mg/m2 over 46-48 hours) IV continuous infusion Repeat every 2 weeks;Cetuximab 500 mg/m2 IV over 2 hours, day 1, every 2 weeks]
  Interventions: Drug: Cetuximab plus FOLFIRI/FOLFOX
- perioperative chemotherapy alone (Active Comparator): FOLFIRI/FOLFOX/CapeOX:routine perioperative chemotherapy including FOLFIRI[Irinotecan 180 mg/m2 IV over 30-90 minutes, day 1 Leucovorin 400 mg/m2 IV infusion to match duration of irinotecan infusion, day 1 5-FU 400 mg/m2 IV bolus day 1, then 1200 mg/m2/day x 2 days (total 2400 mg/m2 over 46-48 hours) continuous infusion Repeat every 2 weeks] or FOLFOX[Oxaliplatin 85 mg/m2 IV over 2 hours, day 1;Leucovorin 400 mg/m2 IV over 2 hours, day 1 5-FU 400 mg/m2 IV bolus on day 1, then 1200 mg/m2/day x 2 days (total 2400 mg/m2 over 46-48 hours) IV continuous infusion Repeat every 2 weeks] or CapeOX[Oxaliplatin 130 mg/m2 IV over 2 hours, day 1 Capecitabine 850-1000mg/m2 twice daily PO for 14 days Repeat every 3 weeks] was adopted in this control arm.
  Interventions: Drug: FOLFIRI/FOLFOX/CapeOX

INTERVENTIONS:
Drug: Cetuximab plus FOLFIRI/FOLFOX — cetuximab was added into the routine perioperative chemotherapy(FOLFIRI/FOLFOX) to evaluate its safety and efficacy
  Other Names: Erbitux; C225
  Arms: chemotherapy plus cetuximab
Drug: FOLFIRI/FOLFOX/CapeOX — to evaluate its safety and efficacy of routine perioperative chemotherapy(FOLFIRI/FOLFOX/CapeOX)
  Other Names: XELOX
  Arms: perioperative chemotherapy alone

SUMMARY:
This study was designed to analyze the prognosis and recurrence predictive factors of high risk patients (Clinical Risk Score≥3) of resectable colorectal liver metastasis.

The efficacy of perioperative chemotherapy plus cetuximab and chemotherapy alone was compared for these patients.

DETAILED DESCRIPTION:
Resection could prolong the survival of colorectal liver metastasis patients, however,the curative resection rate was still low and more than 2/3 of the patients would experience tumor recurrence.This study was designed to formulate a more accurate and individual evaluation system via the multivariate analysis.

Up to now, there was no data to demonstrate the addition of cetuximab to perioperative chemotherapy could decrease recurrence and prolong survival for RAS wild-type, high risk(Clinical Risk Score≥3) resectable colorectal liver metastasis patients. This study was also designed to elucidate this question and to observe the objective response rate(ORR) and the safety data of the regime.

ELIGIBILITY:
Inclusion Criteria:

* good performance status
* pathologic diagnosis of colorectal cancer
* Rat sarcoma viral oncogene homolog(RAS) wild-type
* radiologic confirmation the resectability of liver metastases
* enough future liver remnant
* Clinical Risk Score≥3
* treatment naive
* extra-hepatic metastases could be resected completely, if exist

Exclusion Criteria:

* poor performance status, could not tolerate chemotherapy or operation
* other malignancy history or synchronously
* extra-hepatic metastases could not be resected completely, if exist
* received other treatment previously

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2016-01; Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
disease free survival | From date of hepatectomy until the date of first documented recurrence or metastasis or date of death from any cause, whichever came first, assessed up to 60 months
  months the patient lived from the date of liver resection to the date of disease recurrence or metastasis

SECONDARY OUTCOMES:
overall survival | From date of hepatectomy until the date of first documented death from any cause or the last follow-up if no death happened, assessed up to 60 months
  months the patient lived from the date of liver resection to the date of patient death
objective response rate | from the date of the first chemotherapy until the date two weeks after the completion of the last preoperative chemotherapy, assessed up to 6 weeks
  percent of the number of patients who showed partial response(PR) or complete response(CR) who received preoperative chemotherapy to the number of all the patients enrolled.

CONTACTS AND LOCATIONS:
Overall Officials: Baocai Xing, MD, Study Director — Beijing Cancer Hospital,Peking University
Locations (4):
- China (4):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Primrose J, Falk S, Finch-Jones M, Valle J, O'Reilly D, Siriwardena A, Hornbuckle J, Peterson M, Rees M, Iveson T, Hickish T, Butler R, Stanton L, Dixon E, Little L, Bowers M, Pugh S, Garden OJ, Cunningham D, Maughan T, Bridgewater J. Systemic chemotherapy with or without cetuximab in patients with resectable colorectal liver metastasis: the New EPOC randomised controlled trial. Lancet Oncol. 2014 May;15(6):601-11. doi: 10.1016/S1470-2045(14)70105-6. Epub 2014 Apr 7. PMID 24717919
- [Result] Fong Y, Fortner J, Sun RL, Brennan MF, Blumgart LH. Clinical score for predicting recurrence after hepatic resection for metastatic colorectal cancer: analysis of 1001 consecutive cases. Ann Surg. 1999 Sep;230(3):309-18; discussion 318-21. doi: 10.1097/00000658-199909000-00004. PMID 10493478
- See also: test link — http://ncbi.nlm.nih.gov